CLINICAL TRIAL: NCT04195854
Title: STARS-R Registry: A Retrospective Observational Registry Evaluating the Use of P4HB Scaffolds for Soft Tissue Support in Plastic And Reconstructive Surgery
Brief Title: STARS-R Registry: Retrospective Analysis of Poly-4-hydroxybutyrate (P4HB) Scaffold Use
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Collaborators: Tepha, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1060
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Plastic Surgery; Reconstructive Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: P4HB product — Retrospective use of P4HB in various anatomies

SUMMARY:
This is a retrospective chart review performed at multiple clinics aimed at providing real-world evidence of the use and safety of the P4HB scaffold. Data on patient demographics, relevant medical history, product and procedure used, product safety, and outcome measures will be collected as available.

DETAILED DESCRIPTION:
This is a retrospective chart review performed at multiple clinics aimed at providing real-world evidence of the use and safety of P4HB products. Adults greater than or equal to 18 years old who have undergone a plastic or reconstructive surgical procedure with P4HB on or after January 1, 2014, will be identified using the centers' medical records. Data on patient demographics, relevant medical history, product and procedure used, product safety, and subjective and objective outcome measures will be collected. The data may be used in publication and education and may inform future product development including future clinical trials. The trial will include all consecutive participants who meet inclusion/exclusion criteria with the goal of having up to 5000 participants. A screening log will be kept at the site of all participants screened regardless of whether or not they were included in the analysis. Participants will be entered into the database based on the consecutive group meeting enrollment criteria.

The overall purpose of this study is to gain an understanding of the use and safety of treatments on a historic collection basis. Hypothesis testing is not necessary for the statistical analyses of the generated data. Broad inclusion criteria with few exclusion criteria are utilized so as to avoid censoring historic real-world use of the device.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Underwent plastic or reconstructive surgical procedure with P4HB on or after January 1, 2014 until the date of site initiated data collection
* At least 1 visit of documented post-procedure follow-up

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients greater than or equal to 18 years of age who underwent plastic or reconstructive surgical procedure with P4HB on or after January 1, 2014 until the date of site initiated data collection and who have at least 1 visit of documented post-procedure follow-up
Sampling Method: Non-Probability Sample
Enrollment: 1183 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Real-world utilization of P4HB scaffold | Anticipated 18 months
  To obtain data from real-world utilization of P4HB scaffolds in order to evaluate how and why these products are being used and to assess the safety of these products

SECONDARY OUTCOMES:
Surgeon/patient satisfaction | Anticipated 18 months
  To evaluate surgeon/patient satisfaction with the P4HB scaffold

OTHER OUTCOMES:
Use of Product | Anticipated 18 months
  Type of procedure, reason for procedure, surgical approach tissue assessment, use of other medical devices, concomitant procedures, use of fat grafting
Safety - adverse and serious adverse events | Anticipated 18 months
  Adverse events and serious adverse events related to the study device or procedure, or occurring at procedure anatomy. Medications used in treatment of adverse events
Follow up visits | Anticipated 18 months
  Assessment of healing, menopausal status, Weight, BMI

CONTACTS AND LOCATIONS:
Overall Officials: K Doyle, Study Director — Tepha, Inc/Galatea Surgical
Locations (10):
- United States (10):
  - Aesthetx, Campbell, California
  - Aesthetic Plastic Surgical Institute, Laguna Beach, California
  - Revalla Plastic Surgery and Medical Aesthetics, Littleton, Colorado
  - Sarasota Plastic Surgery, Sarasota, Florida
  - Politis Plastic Surgery, Tampa, Florida
  - Southern Plastic Surgery, Duluth, Georgia
  - Meridian Plastic Surgery, Indianapolis, Indiana
  - Belcara Health, Baltimore, Maryland
  - HKB Cosmetic Surgery, Huntersville, North Carolina
  - Park Cities Surgery, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No